CLINICAL TRIAL: NCT05583422
Title: Evaluating the Uptake and Impact of a Pharmacogenetic Testing Panel in Patients Suspected to be at Increased Risk for Pharmacogenetics-related AEs While Receiving Fluoropyrimidine or Irinotecan Therapy
Brief Title: Evaluating a Pharmacogenetic Testing Panel in Patients Suspected to be at Increased Risk for Pharmacogenetics-related AEs While Receiving Fluoropyrimidine or Irinotecan Therapy
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2022.062; HUM00213709 (Other: University of Michigan)
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: DPYD; UGT1A1
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Cases: This arm will be compiled of prospectively recruited cases for confirmatory testing based on their suspected genotype per Michigan Genomics Initiative and patients who have been retrospectively identified as any patient who had clinical genotype testing and had a variant that was their clinician used to guide the chemotherapy treatment. Prospective patients will undergo confirmatory genetic testing by a CLIA lab and those results will be provided to the patients clinical team at that time.
  Interventions: Genetic: DPYD or UGT1A1 variants
- Controls: This arm will be compiled of all retrospective patients where genetic information was not known prior to receiving treatment.

INTERVENTIONS:
Genetic: DPYD or UGT1A1 variants — any CLIA certified lab can be used for confirmatory testing after patients have been identified through Michigan Genomics Initiative (MGI)
  Groups: Cases

SUMMARY:
This study will be evaluating patients suspected to carry DPYD or UGT1A1 variants based off of Michigan Genomics Initiative (MGI) results. Standard of care treatment will be initiated with either Fluoropyrimidine or Irinotecan therapy. Retrospective collection of treatment related AEs and SAEs, dose delays, dose reductions, and treatment discontinuations will be completed.

DETAILED DESCRIPTION:
Trial was registered as interventional as patients could be enrolled prospectively or retrospectively. Based on data received 2/3/2025, all 16 enrolled cases ended up being identified retrospectively. As the study is now considered to be only retrospective, the record has been updated as not an applicable clinical trial (ACT).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Prospectively enrolled cases:

A. Suspected to carry an actionable DPYD phenotype per MGI and initiating treatment with systemic FP OR suspected to carry an actionable UGT1A1 phenotype per MGI and initiating treatment with irinotecan for cancer

B. The ability to understand and the willingness to sign a written informed consent.

* Retrospective cases:

A. Confirmed actionable DPYD phenotype before treatment with systemic FP OR confirmed actionable UGT1A1 phenotype before treatment with irinotecan

B. Clinician initiated dose reduction of the fluoropyrimidine or irinotecan therapy based upon genotype result

* Retrospective controls:

A. Suspected actionable DPYD phenotype per MGI and treatment with systemic FP OR suspected actionable UGT1A1 phenotype per MGI and treatment with irinotecan

Exclusion Criteria:

* For prospective cases, prior treatment with systemic FP if suspected to carry an actionable DPYD phenotype
* For prospective cases, prior treatment with irinotecan if suspected to carry an actionable UGT1A1 phenotype
* For prospective cases, inability to understand consent or make health-related decisions
* History of allogeneic bone marrow transplant prior to genotype testing
* History of liver transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have been retrospectively identified as any patient who had clinical genotype testing and had a variant that was their clinician used to guide the chemotherapy treatment.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Comparison of grade 3 or higher AEs and SAEs | five months from treatment initiation
  Compare rates of grade 3 or higher AEs and SAEs to fluoropyrimidine or irinotecan treatment between subjects with confirmed DPYD or UGT1A1 variants before chemotherapy treatment to retrospective matched controls without confirmatory PGx testing

SECONDARY OUTCOMES:
Comparison of PGx genotypes to MGI genotypes | five months from treatment initiation
  clinical genotypes and MGI genotypes for participants will be considered concordant if they identify the same DPYD or UGT1A1 variant and discordant if they do not
Comparison of rates of dose reductions | five months from treatment initiation
  A decrease in dose of standard of care treatment by >10% of the dose administered for the prior cycle
Comparison of treatment cycle delays | five months from treatment initiation
  Any prolongation of the initiation of the following scheduled treatment cycle due to toxicity as documented by the patient's medical team
Comparison of treatment discontinuation | five months from treatment initiation
  Any discontinuation due to clinician-documented toxicity
Clinician acceptance of supportive care pharmacogenetics | 6 months post first standard of care treatment
  Evaluation of the amount of new prescriptions written with identified genetic interactions

CONTACTS AND LOCATIONS:
Overall Officials: Amy Pasternak, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No